CLINICAL TRIAL: NCT02990494
Title: Prevention & Promotion in the Treatment of Obesity
Acronym: PROSPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Kathryn E. Demos, Assistant Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R03DK106405-01A1 (NIH)
Record Dates: First submitted 2016-12-07; First posted 2016-12-13 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- STANDARD (Active Comparator): 12-week Internet-delivered behavioral weight loss program
  Interventions: Behavioral: STANDARD
- PREVENT (Experimental): an enhanced 12-week Internet-delivered behavioral weight loss program focused on preventing future negative consequences
  Interventions: Behavioral: PREVENT
- PROMOTE (Experimental): an enhanced 12-week Internet-delivered behavioral weight loss program focused on promoting future benefits
  Interventions: Behavioral: PROMOTE

INTERVENTIONS:
Behavioral: STANDARD — Standard Internet-delivered behavioral weight loss
  Other Names: Standard Internet-delivered behavioral weight loss
  Arms: STANDARD
Behavioral: PREVENT — enhanced standard Internet-delivered behavioral weight loss program
  Other Names: PREVENT Internet-delivered behavioral weight loss
  Arms: PREVENT
Behavioral: PROMOTE — enhanced standard Internet-delivered behavioral weight loss program
  Other Names: PROMOTE Internet-delivered behavioral weight loss
  Arms: PROMOTE

SUMMARY:
Making healthy food choices requires sacrificing immediate pleasures of consuming high calorie foods in order to achieve long-term health goals. Two strategies to encourage such future thinking are 1) focusing on the long-term consequences of consuming unhealthy foods, and 2) focusing on the long-term benefits of avoiding these unhealthy foods. Two novel behavioral weight loss (BWL) interventions will be developed based on these strategies (PREVENT and PROMOTE) and compared to standard Internet-delivered BWL to test their feasibility and efficacy in changing food choice decision-making, reducing food cravings, and ultimate weight loss.

DETAILED DESCRIPTION:
Obesity is one of the most important public health issues today, contributing to many of the primary causes of morbidity and mortality in the United States. Still, treatment remains difficult and many people continually struggle to lose weight. Thus there is critical need for improvements in methods for treating obesity. One potential reason weight control is so difficult is the need to sacrifice immediate pleasures for long-term goals. This requires placing significant value on future outcomes, such as health.

One strategy for doing so is to focus on the potential benefits of avoiding unhealthy choices. Health messaging studies suggest that messages focused on promoting long-term benefits of healthier choices may be effective in encouraging initiation of, or positive attitudes toward, healthy behaviors, however, longer-term effects of these messages have not been studied in the context of obesity. By contrast, behavioral economic work on Prospect Theory suggests focusing on preventing future negative consequences may be superior, and the threat of weight gain is a more powerful motivator than the benefit of weight loss. Although prevention strategies have been successfully employed in smoking cessation and anti-smoking campaigns, they are not typically used in obesity treatment. In promising preliminary neuroimaging work, the investigators identified increases in brain regions involved in inhibitory control and decreases in cravings when using this PREVENT strategy.

The goal of this R03 is to test whether an intervention built upon the goal to PREVENT long-term consequences of weight gain versus an intervention built upon the goal to PROMOTE long-term benefits of weight loss is beneficial in altering valuation of health and taste in food choice decision-making, encouraging adherence, reducing food cravings and consumption, and ultimate weight loss, as compared to a standard behavioral weight loss program (BWL). A total of 90 overweight/obese men and women will be randomly assigned to either PREVENT, PROMOTE, or standard BWL. Each intervention will have one in-person training session wherein participants will learn key strategies of their assigned program, and the remaining 12 weekly lessons will be delivered via internet. Baseline and 3-month (post-treatment) assessments will include the food choice decision-making task featured in the parent K01 to measure valuation of health and taste, weight measurement, and measurement of food cravings and consumption. To address feasibility, adherence and engagement measures (i.e., lessons viewed, self-monitoring) will be collected during the internet program, and memory for lesson content will be assessed post-treatment. Individual difference measures will also be collected to provide preliminary data on factors that may influence success in each arm.

This project tests innovative approaches in the clinical treatment of obesity and will provide new insights into the potential role of prevention versus promotion strategies for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* ages 25-60
* currently overweight or obese (BMI 25-45 kg/m2)

Exclusion Criteria:

* lack of access to a computer and the Internet (needed once per week),
* weight loss medications
* neurological or psychiatric conditions including but not limited to schizophrenia, and bipolar disorder
* inability to attend assessments
* lack of interest in participating in a behavioral weight loss trial
* serious current physical disease for which physician supervision of diet and exercise prescription is needed
* physical problems that limit the ability to exercise
* participation in a weight loss program within the last 2 months
* intention to become pregnant in the next 3 months

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in food choice decision-making task | baseline baseline and within 30 days of intervention conclusion

SECONDARY OUTCOMES:
adherence and acceptability questionnaire | during 12-week intervention and within 30 days of intervention conclusion
  assessing adherence (number of lessons viewed and self-monitoring data entered by participants) throughout the intervention and acceptability of the intervention following treatment
change in cravings and consumption questionnaire | from baseline to within 30 days of intervention conclusion
change in scale-measured body weight | from baseline to within 30 days of intervention conclusion